CLINICAL TRIAL: NCT01292330
Title: A Clinical Study to Evaluate the Clinical Outcomes of Hepatectomy With Nutritional Risk After Preoperative Nutritional Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Dr. Yilei Mao, Peking Union Medical College Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PUMCH-Liver surgery -Nutrition
Record Dates: First submitted 2011-02-06; First posted 2011-02-09 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2011-02

CONDITIONS: Liver Cancer
Keywords: liver Tumor
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: nutritional support before operation — nutritional support before operation for more than 4 days

SUMMARY:
Objective:to Study the clinical outcomes of hepatectomy with Nutritional risk After Preoperative Nutritional Support.

Study design:

1.Prospective，randomized, controlled clinical study;2.Patients: The subjects were from Peking Union Medical College Hospital (PUMCH).

Study arrangement:

1. The collection of patients with selected standard
2. Preoperative evaluation included nutritional status,liver function and tumor characteristics
3. The experimental group received Preoperative Nutritional Support for 4 days,the control group got nothing
4. Both groups received conventional therapy after operation
5. The comparation of the clinical outcomes in both groups

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of hepatocellular carcinoma (HCC) was made before operation
2. Nutritional Risk Screening 2002(NRS-2002) was Greater or equal 3 points with in 24 hours after admission

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-09 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | 2 years
  postoperative complications especially infectious complications

SECONDARY OUTCOMES:
hospitalization expenses and length of stay | 2 years
  hospitalization expenses:nutrition-related expenses length of stay:from the date of the operation to the date of Discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Yilei Mao, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lu X, Li Y, Yang H, Sang X, Zhao H, Xu H, Du S, Xu Y, Chi T, Zhong S, Yu K, Mao Y. Improvement of nutritional support strategies after surgery for benign liver tumor through nutritional risk screening: a prospective, randomized, controlled, single-blind clinical study. Hepatobiliary Surg Nutr. 2013 Feb;2(1):14-21. doi: 10.3978/j.issn.2304-3881.2012.11.04. PMID 24570910